CLINICAL TRIAL: NCT03468231
Title: Sorafenib Plus Hepatic Artery Infusion Chemotherapy of Oxaliplatin, Fluorouracil/Leucovorin Versus Sorafenib Plus Hepatic Artery Infusion Chemotherapy of Oxaliplatin for Hepatocellular Carcinoma With Major Portal Vein Tumor Thrombosis
Brief Title: HAIC of FOLFOX vs. HAIC of OXA for Advanced HCC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); Dongguan People's Hospital (Other Government); Kaiping Central Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Guangzhou No.12 People's Hospital (Other Government); The First Affiliated Hospital of University of South China (Other)
Responsible Party: Principal Investigator, Shi Ming, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HCC-20180309
Record Dates: First submitted 2018-03-11; First posted 2018-03-16 (Actual); Last update posted 2018-03-16 (Actual); Status verified 2018-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Hepatic arterial infusion chemotherapy; Sorafenib; Oxaliplatin plus Fluorouracil/Leucovorin; Oxaliplatin
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib; Oxaliplatin; Fluorouracil; Leucovorin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: In the OXA group, saline replace the fluorouracil and leucovorin solution and patients are treated the same time as the FOLFOX group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sorafenib plus HAIC of FOLFOX (Active Comparator): Sorafenib combined with Hepatic arterial infusion chemotherapy with Oxaliplatin, Fluorouracil and Leucovorin
  Interventions: Drug: Sorafenib; Drug: HAIC of FOLFOX
- Sorafenbi plus HAIC of OXA (Experimental): Sorafenib combined with Hepatic arterial infusion chemotherapy with Oxaliplatin
  Interventions: Drug: Sorafenib; Drug: HAIC of OXA

INTERVENTIONS:
Drug: Sorafenib — Oral Sorafenib, 400mg, Bid
Drug: HAIC of FOLFOX — administration of Oxaliplatin , fluorouracil, and leucovorin via the tumor feeding arteries
  Other Names: Oxaliplatin , fluorouracil, and leucovorin
  Arms: Sorafenib plus HAIC of FOLFOX
Drug: HAIC of OXA — administration of Oxaliplatin via the tumor feeding arteries
  Other Names: Oxaliplatin
  Arms: Sorafenbi plus HAIC of OXA

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of hepatic arterial infusion chemotherapy (HAIC) of oxaliplatin plus fluorouracil/leucovorin compared with HAIC of oxaliplatin alone in patients with hepatocellular carcinoma (HCC) with major portal venous tumor thrombus (PVTT).

DETAILED DESCRIPTION:
Sorafenib is the most widely used palliative treatment for hepatocellular carcinoma (HCC) patients with portal venous tumor thrombus (PVTT). Our previous prospective study revealed that sorafenib combined with hepatic arterial infusion chemotherapy (HAIC) of oxaliplatin plus fluorouracil/leucovorin confer a survival benefit to HCC with major PVTT. However, HAIC of fluorouracil is not such for advanced HCC. Whether HAIC of oxaliplatin is as effective as HAIC of oxaliplatin plus fluorouracil/leucovorin is controversial. Thus, the investigators carried out this prospective randomized control study to find out it.

ELIGIBILITY:
Inclusion Criteria:

The diagnosis of HCC was based on the diagnostic criteria for HCC used by the European Association for the Study of the Liver (EASL)

* Patients must have at least one tumor lesion that can be accurately measured according to EASL criteria.
* diagnosed with major or main portal vein invasion (Vp3 or Vp4)
* KPS≥70；
* with no previous treatment
* No Cirrhosis or cirrhotic status of Child-Pugh class A only
* Not amendable to surgical resection ,local ablative therapy and any other cured treatment.
* The following laboratory parameters:
* Platelet count ≥ 75,000/µL
* Hemoglobin ≥ 8.5 g/dL
* Total bilirubin ≤ 30mmol/L
* Serum albumin ≥ 30 g/L
* ASL and AST ≤ 5 x upper limit of normal
* Serum creatinine ≤ 1.5 x upper limit of normal
* INR ≤ 1.5 or PT/APTT within normal limits
* Absolute neutrophil count (ANC) >1,500/mm3
* Ability to understand the protocol and to agree to and sign a written informed consent document

Exclusion Criteria:

* Evidence of hepatic decompensation including ascites, gastrointestinal bleeding or hepatic encephalopathy
* Known history of HIV
* History of organ allograft
* Known or suspected allergy to the investigational agents or any agent given in association with this trial.
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* Evidence of bleeding diathesis.
* Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry.
* Any other hemorrhage/bleeding event > CTCAE Grade 3 within 4 weeks of first dose of study drug
* Serious non-healing wound, ulcer, or bone fracture
* Known central nervous system tumors including metastatic brain disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2018-03-09 (Actual); Primary Completion 2019-09-09 (Estimated); Study Completion 2020-03-09 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 10 months
  Overall survival

SECONDARY OUTCOMES:
Progress free survival | 10 months
  Progress free survival
Adverse Events | 30 days
  Number of adverse events. Postoperative adverse events were graded based on CTCAE v4.0
Number of of Patients developed Adverse Events | 30 days
  Number of of patients who developed adverse event. Postoperative adverse events were graded based on CTCAE v4.0
Tumor response | 10 months
  overall response

CONTACTS AND LOCATIONS:
Overall Officials: Ming Shi, MD, Principal Investigator — The Department of Hepatobiliary Oncology of Sun Yat-sen University Cancer Center
Locations (7):
- China (7):
  - Dongguan People's Hospital, Dongguan, Guangdong
  - Cancer Center Sun Yat-sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Guangzhou Twelfth People 's Hospital, Guangzhou, Guangdong
  - Kaiping Central Hospital, Kaiping, Guangdong
  - First Affiliated Hospital of University Of South China, Hengyang, Hunan
  - The First Affiliated Hospital Of Xi'an Jiaotong University, Xi’an, Shanxi